# **Cover Page**

**Proposal Title:** Effect of preoperative oral administration of Ibuprofen and Acetaminophen on the anesthetic efficacy of buccal infiltration during vital pulpotomy of mandibular primary molars: A Prospective, Double-blinded, Randomized Controlled Trial

### First Investigator: Reham Khaled Abou El Fadl

Lecturer Pediatric Dentistry, Dental Public Health Department, Faculty of Dentistry, Ain Shams University

MPH Public Health, Imperial College of London

reham.k.abouelfadl@gmail.com

**Second Investigator: Maram Obeid** 

Lecturer Endodontics Department, Faculty of Dentistry, Ain Shams University

maramobeid@icloud.com

### **Introduction:**

Pain is one of the most unpleasant sensations that human beings may experience throughout their lives. Pain control, particularly in children, is a vital part for a successful dental treatment. Optimal pain control measures result in building up trust and facilitate the entire procedure <sup>(1)</sup>.

Effective pain control while delivering dental treatment is considered as the keystone of pediatric behavior management. The mandibular block is the local anesthesia technique of choice when treating mandibular primary or permanent molars. A number of disadvantages, however, have been associated with this technique. The duration of anesthesia makes the uncomfortable numb feeling last long after the end of dental treatment, often resulting in lip or tongue biting <sup>(2)</sup>. Furthermore, triggering a successful mandibular block involves a degree of difficulty rendering the injection stressful for both the clinician and the patient. Thus the administration of the anesthetic agent is still considered the most painful part of most dental procedures <sup>(3)</sup>.

Investigators have tested other techniques where infiltration anesthesia was used successfully to restore maxillary teeth but has been avoided in the mandibular molar regions because of denser bone that does not allow adequate dissemination of the anesthetic <sup>(2)</sup>. Some studies assessed the effectiveness of mandibular infiltration in restoring primary molars in children and concluded that infiltration anesthesia was successful <sup>(4, 5)</sup>.

Generally, pain assessment is very subjective; it can be only indirectly measured in children through verbal self-report or observation of behaviors that suggest pain <sup>(6)</sup>. There are several pain scale indicators that can be used with children, including the FACES pain scale and the Wong-Baker FACES scale <sup>(7,8)</sup>.

Researchers have studied different ways to have better anesthesia in permanent teeth. Premedication with analgesic agents has been proposed as alternatives with controversial results <sup>(9)</sup>. Numerous analgesics are used for pain control ranging from opioids to non-narcotic analgesics including acetaminophen (Flavol) and non-steroidal anti-inflammatory drugs (NSAIDs) (Brufen). NSAIDS block the cyclooxygenase enzyme in the pathway that produces prostaglandins, resulting in lower levels of inflammation-inciting prostaglandins <sup>(10, 11)</sup>. Although the action of acetaminophen is unknown, it has been suggested that it interferes with inflammation by diminishing the synthesis of prostaglandins (possibly PGF2); and also alters the transmission of pain by acting directly on an unknown site in the brain <sup>(12, 13)</sup>.

### **Objective:**

The purpose of this double-blinded, randomized, prospective study will be to determine the effectiveness of buccal infiltration during vital pulpotomy in mandibular primary molars in relation to two different analysesic premedications.

# Methodology

## **Recruitment/Study setting:**

A total of 60 healthy children will be recruited from the outpatient clinic of the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University. One author will screen and recruit all the patients in the study.

### **Inclusion and Exclusion Criteria**

Preoperative periapical radiographs will be obtained for all subjects prior to inclusion in the study and participation will be based on the following eligibility criteria for children:

Of age group 7–9 years

Without systemic or mental disorders.

Who could be categorized as cooperative according to *Wright's classification* for child behavior

Ability of child to understand the use of pain scales;

Having at least one lower second primary molar with deep caries indicated for pulpotomy;

Absence of any periapical or furcation radiolucency on radiographs,

Absence of any signs of internal or external resorption on radiographs,

A vital coronal pulp on access opening.

Exclusion criteria include any allergic reactions, sensitivity, or contraindications to any tested drugs or history of bleeding problems. Patients who had taken analgesics within 12 hours before administration of the study drugs or those having active pain, pulpitis or abscess related to the designated mandibular molar will not be included. Children with special health care needs or any systemic problems will be excluded from our study as well.

### **Ethical Considerations:**

Patients who failed to fulfill the eligibility criteria of the study will receive any necessary dental treatment in the outpatient clinic. Parents of eligible children will be informed about the nature of the procedure, the purpose of the study, any possible discomfort or risks and a signed informed consent will be obtained from them prior to enrollment.

### **Interventions:**

Subjects meeting the inclusion criteria will be divided into three groups (24 patients/group) and will be given one of the following three drugs:

- Brufen syrup (Ibuprofen BP 100 mg/5 ml, an orange-coloured, orange-flavoured, syrupy suspension)
- Fevano Syrup (Paracetamol 200 mg/5ml. an orange-coloured, mango flavoured)
- Sansovit Iron (Multivitamin +Iron, an orange-coloured, orange-flavoured) as a control

All solutions will be placed in medicine bottles and will be randomly assigned 3-digit numbers by one of the authors to ensure blinding. To ensure randomization and allocation concealment, children will be randomly assigned to the three groups using computer-generated numbers. The numbers of patients in each group will be written on paper which will be then kept in a sealed opaque envelope. Each child will be asked to choose one of the envelopes and thus assignment to one of the three groups will be based on the chosen number.

Each child will then receive an age-dosed volume of the assigned drug 1 hour before starting the treatment. Before taking the drug, the patients will be asked to rate their pain using **Wong Baker FACES** pain assessment tool. For all subjects, the anesthetic solution will be 4% Articaine with adrenaline 1:200 000. Topical anesthesia will be applied for 2-3 min on previously dried mucosa before administration of the solution. The solution will be injected by the same clinician by using self-aspirating syringes and 27 gauge, short needles.

Children will be asked about lip numbness every 3 minutes for 10 minutes. Ten minutes after injection, removal of caries and coronal access will be performed. Patients will be asked to rate any pain felt during treatment using the same assessment tool.

A pilot study will be conducted in a group of 10 children to assess for feasibility and success of combining buccal infiltration with the tested analgesic premeditations.

### **References:**

- 1. Walton RE, Reader A, Nusstein JM (2008). Local anesthesia. In: Torabinejad M, Walton RE, eds. Endodontics, Principles and Practice. 4th ed. St Louis, MO: Saunders Elsevier pp. 129–47
- 2. Oulis CJ, Vadiakas GP, Vasilopoulou A. The effectiveness of mandibular infiltration compared to mandibular block anesthesia in treating primary molars in children. Pediatric dentistry 1996; 18:301-5.

- 3. Fiset L, Milgrom P, Weinstein P, Getz T, Glassman P. Psychophysiological responses to dental injections. J Am Dent Assoc. 1985; 111:578–82.
- 4. Dudkiewicz A, Schwartz S, Lalibert6 R: Effectiveness of mandibular infiltration in children using the local anesthetic Ultracaine (articaine hydrochloride). Can Dent Assoc 53:29-31, 1987.
- 5. Wright GZ, Weinberger SJ, Marti R, Plotzke O: The effectiveness of infiltration anesthesia in the mandibular primary molar region. Pediatr Dent 13:278-83, 1991
- 6. Schechter NL, Berde CB, Yaster M, Eds: Pain in Infants, Children, and Adolescents. Baltimore: Williams and Wilkins, 1993, pp 3-11
- 7. Barrêtto EPR, Ferreira EF, Pordeus IA. Evaluation of toothache severity in children using a visual analog scale of faces. Pediatr Dent 2004;26(6):485-91.
- 8. Hicks CL, von Baeyer CL, Spafford P, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: Toward a common metric in pediatric pain measurement. Pain 2001;93(2):173-83.
- 9. Modaresi J, Dianat O, Mozayeni MA (2006). The efficacy comparison of ibuprofen, acetaminophen-codeine, and placebo premedication therapy on the depth of anesthesia during treatment of inflamed teeth. Oral Surg.102:399–403.
- 10. Trowbridge H, Emling R. Chemical mediators of the vascular response. In: Trowbridge H, Emling R, eds. Inflammation: a review of the process, 5th ed. Chicago: Quintessence Publishing Co., 1997:33.
- 11. Wynn R, Meiller T, Crossley H. Drug information handbook for dentistry, 9th ed. Hudson: Lexi-Comp, 2003:356.
- 12. Ingle JI, Walton RE, Malamed SF, et al. Preparation for endodontic treatment. In: Ingle JI, Bakland LK, eds. Endodontics, 5th ed. Hamilton: BC Decker, 2002;385.
- 13. Malamed SF. Management of pain and anxiety. In: Cohen S, Burns R, eds. Pathways of the pulp, 8th ed. St. Louis: Mosby, 2002;735–7.